CLINICAL TRIAL: NCT02142634
Title: Randomised, Double-blind, Placebo-controlled, Multi-centre Trial on the Efficacy and Safety of Budesonide for Induction of Remission in Incomplete Microscopic Colitis
Brief Title: Budesonide for Induction of Remission in Incomplete Microscopic Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUG-3/MIC; 2013-001912-31 (EudraCT Number)
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Incomplete Microscopic Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Budesonide granules 9 mg
  Interventions: Drug: Budesonide granules 9 mg
- B (Placebo Comparator): Placebo granules
  Interventions: Drug: Placebo granules

INTERVENTIONS:
Drug: Budesonide granules 9 mg — per day
  Arms: A
Drug: Placebo granules — per day
  Arms: B

SUMMARY:
The purpose of this study is to demonstrate the efficacy of budesonide for the treatment of active incomplete microscopic colitis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically established diagnosis of incomplete microscopic colitis (MCi)
* History of chronic non-bloody, watery diarrhoea
* Clinically active disease

Exclusion Criteria:

* Other significant abnormalities in colonoscopy
* Infectious cause of diarrhoea
* Clinical suspicion of drug-induced diarrhoea
* Prior and present MC
* History of bowel resection
* Radiation therapy of the abdominal or pelvic region
* Positive antibody titres for celiac disease
* Untreated active thyroid dysfunction
* Any severe concomitant cardiovascular, renal, endocrine, or psychiatric disorder reducing life expectancy
* Abnormal hepatic function
* Tuberculosis, hypertension, diabetes mellitus, osteoporosis, peptic ulcer disease, glaucoma, cataract, or infection if careful medical monitoring is not ensured
* History of colorectal cancer
* History of cancer (other than colorectal) in the last 5 years
* Therapy with immunomodulators/budesonide or other steroids/antibiotics/anti-diarrhoeal drugs
* Current or intended pregnancy or breast-feeding
* Doubt about the patient's cooperation, e.g. because of addiction to alcohol or drugs
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission | 8 weeks

SECONDARY OUTCOMES:
Rate of clinical remission | 2 weeks
Rate of clinical remission | 6 weeks
Time to remission | 8 weeks
Number of formed/soft/watery stools per week | 8 weeks
Number of days with abdominal pain | 8 weeks
Number of days with urgency | 8 weeks
Rate of histological remission | 8 weeks
Physician's global assessment at final visit | 8 weeks
Quality of life | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Münch, MD, Principal Investigator — University Hospital of Linköping, Dept. of Gastroenterology and Hepatology
Locations (2):
- Centre for Digestive Diseases, Hamburg, Germany
- University Hospital of Linköping, Dept. of Gastroenterology and Hepatology, Linköping, Sweden